CLINICAL TRIAL: NCT03194958
Title: Helping the Poor Quit Smoking: Specialized Quitlines and Meeting Basic Needs
Brief Title: Helping Poor Smokers Quit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Matthew Kreuter, Associate Dean for Public Health; Director, Washington University School of Medicine
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Health Services Research
Other Study IDs: R01CA201429 (NIH); R01CA201429 (NIH)
Record Dates: First submitted 2017-06-19; First posted 2017-06-21 (Actual); Results first posted 2023-12-26 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Smoking Cessation; Smoking, Tobacco; Smoking, Cigarette; Smoking, Pipe; Smoking (Tobacco) Addiction; Smoking; Tobacco Use; Tobacco Dependence; Tobacco Use Cessation; Tobacco Smoking; Tobacco; Use, Rehabilitation; Nicotine Dependence; Nicotine Use Disorder; Nicotine Dependence, Cigarettes; Nicotine Dependence Tobacco Product
MeSH Terms: conditions — Smoking Cessation; Tobacco Smoking; Cigarette Smoking; Pipe Smoking; Smoking; Behavior, Addictive; Tobacco Use; Tobacco Use Disorder; Tobacco Use Cessation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Standard Quitline (No Intervention): Participants will receive standard Missouri quitline services
- Specialized Quitline (Experimental): Participants will receive an enhanced version of the standard quitline services
  Interventions: Behavioral: Specialized Quitline
- Standard Quitline with Basic Needs Navigator (Experimental): Participants receive standard quitline services with navigator
  Interventions: Behavioral: Basic Needs Navigator
- Specialized Quitline with Basic Needs Navigator (Experimental): Participants receive enhanced quitline services with navigator
  Interventions: Behavioral: Specialized Quitline; Behavioral: Basic Needs Navigator

INTERVENTIONS:
Behavioral: Specialized Quitline — Very low-income smokers are different from other smokers in important ways not always addressed by standard quitline services. The research team and Alere staff has created custom protocols, scripts, prompts and other content to maximize intervention relevance and acceptability to very low-income smokers. Research Implementation Unit (RIU) coaches who will be delivering the Specialized Quitline services have received training from clinical quitline staff, the research team and 2-1-1 staff who have extensive experience with the target population. Focus areas for training and distinctive content and protocol for the Specialized Quitline include: health literacy, abstract vs. concrete language, lived experience, resource constraints, future orientation, getting cigarettes, living situation, phone/internet access.
  Arms: Specialized Quitline; Specialized Quitline with Basic Needs Navigator
Behavioral: Basic Needs Navigator — Navigators will: (1) identify and assess smokers' needs, including the reasons they called 2-1-1; (2) jointly generate solutions to address the needs; (3) develop plans to carry out the solutions, including; (4) help prioritize among multiple needs; (5) identify community resources that could help solve the problem; (6) determine eligibility for services; (7) help smokers access available resources by scheduling appointments and provide appointment reminders; (8) prepare smokers to interact with service agencies and/or act as an advocate on their behalf; (9) provide instrumental support such as arranging transportation; (10) actively intervene to resolve barriers to basic needs solutions; (11) oversee follow-up of problem solving actions; and (12) review progress made towards resolving unmet basic needs and adapt solutions accordingly.
  Arms: Specialized Quitline with Basic Needs Navigator; Standard Quitline with Basic Needs Navigator

SUMMARY:
Using a 2x2 randomized factorial design, we will conduct a statewide field trial in Missouri to compare the relative and combined effects of these two strategies for augmenting an existing, evidence-based tobacco quitline program. Among 2000 low-income smokers, half will receive standard Missouri quitline services and half will receive new Specialized Quitline services targeted to this group. In each of these groups, half also will receive calls from a trained navigator to help them address unmet Basic Needs and the accompanying psychological distress that act as barriers to smoking cessation.

DETAILED DESCRIPTION:
2-1-1 information specialists will deliver standard service, then ask a random number of callers per day if they would be willing to answer a few health questions as part of a new 2-1-1 service. Callers eligible to receive the invitation to screen for study eligibility will be: Missouri residents, calling for themselves, English-speaking, and not in acute crisis. Eligible smokers will then be asked if they are willing to share their contact information with a research team conducting a study to help smokers quit. Smokers who agree to share their contact information will be considered "enrolled". Trained 2-1-1 operators will record all recruitment screening data in a secure electronic database that is shared with research staff. Research staff will attempt to reach enrolled smokers by phone by the next business day.

Alere, through the Missouri Tobacco Quitline, will provide quitline services to smokers in all study conditions. Contact information and study group assignment for smokers will be provided to Alere via secure data transfer.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Missouri resident
* English speaking
* Not in crisis
* Smoke cigarettes every day of the week
* Planning to quit smoking in the next 30 days
* Comfortable receiving calls from smoking expert and project team
* Willing to provide phone numbers to be reached

Exclusion Criteria:

* Pregnant or planning to become pregnant in the next 3 months
* Currently breastfeeding
* Insurance through employer
* Currently enrolled in smoking quitline

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1944 (Actual)
Dates: Start 2017-06-05 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Kreuter, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University in St. Louis, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Boyum S, Kreuter MW, McQueen A, Thompson T, Greer R. Getting help from 2-1-1: A statewide study of referral outcomes. J Soc Serv Res. 2016;42(3):402-411. doi: 10.1080/01488376.2015.1109576. Epub 2016 Jan 22. PMID 28260823
- [Background] Cappelletti ER, Kreuter MW, Boyum S, Thompson T. Basic needs, stress and the effects of tailored health communication in vulnerable populations. Health Educ Res. 2015 Aug;30(4):591-8. doi: 10.1093/her/cyv033. PMID 26187910
- [Background] Kreuter MW, McQueen A, Boyum S, Fu Q. Unmet basic needs and health intervention effectiveness in low-income populations. Prev Med. 2016 Oct;91:70-75. doi: 10.1016/j.ypmed.2016.08.006. Epub 2016 Aug 3. PMID 27496395
- [Background] Thompson T, Kreuter MW, Boyum S. Promoting Health by Addressing Basic Needs: Effect of Problem Resolution on Contacting Health Referrals. Health Educ Behav. 2016 Apr;43(2):201-7. doi: 10.1177/1090198115599396. Epub 2015 Aug 20. PMID 26293458
- [Background] Zanis DA, Hollm RE, Derr D, Ibrahim JK, Collins BN, Coviello D, Melochick JR. Comparing intervention strategies among rural, low SES, young adult tobacco users. Am J Health Behav. 2011 Mar-Apr;35(2):240-7. doi: 10.5993/ajhb.35.2.11. PMID 21204686
- [Background] Richter KP, Shireman TI, Ellerbeck EF, Cupertino AP, Catley D, Cox LS, Preacher KJ, Spaulding R, Mussulman LM, Nazir N, Hunt JJ, Lambart L. Comparative and cost effectiveness of telemedicine versus telephone counseling for smoking cessation. J Med Internet Res. 2015 May 8;17(5):e113. doi: 10.2196/jmir.3975. PMID 25956257
- [Background] Ferketich AK, Pennell M, Seiber EE, Wang L, Farietta T, Jin Y, Wewers ME. Provider-delivered tobacco dependence treatment to Medicaid smokers. Nicotine Tob Res. 2014 Jun;16(6):786-93. doi: 10.1093/ntr/ntt221. Epub 2014 Jan 28. PMID 24474305
- [Background] Bush T, Levine MD, Beebe LA, Cerutti B, Deprey M, McAfee T, Boeckman L, Zbikowski S. Addressing weight gain in smoking cessation treatment: a randomized controlled trial. Am J Health Promot. 2012 Nov-Dec;27(2):94-102. doi: 10.4278/ajhp.110603-QUAN-238. PMID 23113779
- [Background] Smith SS, Keller PA, Kobinsky KH, Baker TB, Fraser DL, Bush T, Magnusson B, Zbikowski SM, McAfee TA, Fiore MC. Enhancing tobacco quitline effectiveness: identifying a superior pharmacotherapy adjuvant. Nicotine Tob Res. 2013 Mar;15(3):718-28. doi: 10.1093/ntr/nts186. Epub 2012 Sep 19. PMID 22992296
- [Background] Perry RJ, Keller PA, Fraser D, Fiore MC. Fax to quit: a model for delivery of tobacco cessation services to Wisconsin residents. WMJ. 2005 May;104(4):37-40, 44. PMID 16117232
- [Background] Stead LF, Perera R, Lancaster T. Telephone counselling for smoking cessation. Cochrane Database Syst Rev. 2006 Jul 19;(3):CD002850. doi: 10.1002/14651858.CD002850.pub2. PMID 16855992
- [Background] Fiore MC. US public health service clinical practice guideline: treating tobacco use and dependence. Respir Care. 2000 Oct;45(10):1200-62. PMID 11054899
- [Background] Stead LF, Buitrago D, Preciado N, Sanchez G, Hartmann-Boyce J, Lancaster T. Physician advice for smoking cessation. Cochrane Database Syst Rev. 2013 May 31;2013(5):CD000165. doi: 10.1002/14651858.CD000165.pub4. PMID 23728631
- [Background] Bryant J, Bonevski B, Paul C, McElduff P, Attia J. A systematic review and meta-analysis of the effectiveness of behavioural smoking cessation interventions in selected disadvantaged groups. Addiction. 2011 Sep;106(9):1568-85. doi: 10.1111/j.1360-0443.2011.03467.x. Epub 2011 Jul 22. PMID 21489007
- [Background] Lichtenstein E, Glasgow RE, Lando HA, Ossip-Klein DJ, Boles SM. Telephone counseling for smoking cessation: rationales and meta-analytic review of evidence. Health Educ Res. 1996 Jun;11(2):243-57. doi: 10.1093/her/11.2.243. PMID 10163409
- [Background] Stead LF, Lancaster T, Perera R. Telephone counselling for smoking cessation. Cochrane Database Syst Rev. 2003;(1):CD002850. doi: 10.1002/14651858.CD002850. PMID 12535442
- [Background] Kreuter MW, Eddens KS, Alcaraz KI, Rath S, Lai C, Caito N, Greer R, Bridges N, Purnell JQ, Wells A, Fu Q, Walsh C, Eckstein E, Griffith J, Nelson A, Paine C, Aziz T, Roux AM. Use of cancer control referrals by 2-1-1 callers: a randomized trial. Am J Prev Med. 2012 Dec;43(6 Suppl 5):S425-34. doi: 10.1016/j.amepre.2012.09.004. PMID 23157761
- [Background] Agaku IT, King BA, Dube SR; Centers for Disease Control and Prevention (CDC). Current cigarette smoking among adults - United States, 2005-2012. MMWR Morb Mortal Wkly Rep. 2014 Jan 17;63(2):29-34. PMID 24430098
- [Background] Siahpush M, McNeill A, Borland R, Fong GT. Socioeconomic variations in nicotine dependence, self-efficacy, and intention to quit across four countries: findings from the International Tobacco Control (ITC) Four Country Survey. Tob Control. 2006 Jun;15 Suppl 3(Suppl 3):iii71-5. doi: 10.1136/tc.2004.008763. PMID 16754950
- [Background] Barbeau EM, Krieger N, Soobader MJ. Working class matters: socioeconomic disadvantage, race/ethnicity, gender, and smoking in NHIS 2000. Am J Public Health. 2004 Feb;94(2):269-78. doi: 10.2105/ajph.94.2.269. PMID 14759942
- [Background] Flint AJ, Novotny TE. Poverty status and cigarette smoking prevalence and cessation in the United States, 1983-1993: the independent risk of being poor. Tob Control. 1997 Spring;6(1):14-8. doi: 10.1136/tc.6.1.14. PMID 9176981
- [Background] Businelle MS, Kendzor DE, Reitzel LR, Costello TJ, Cofta-Woerpel L, Li Y, Mazas CA, Vidrine JI, Cinciripini PM, Greisinger AJ, Wetter DW. Mechanisms linking socioeconomic status to smoking cessation: a structural equation modeling approach. Health Psychol. 2010 May;29(3):262-73. doi: 10.1037/a0019285. PMID 20496980
- [Background] Reid JL, Hammond D, Boudreau C, Fong GT, Siahpush M; ITC Collaboration. Socioeconomic disparities in quit intentions, quit attempts, and smoking abstinence among smokers in four western countries: findings from the International Tobacco Control Four Country Survey. Nicotine Tob Res. 2010 Oct;12 Suppl(Suppl 1):S20-33. doi: 10.1093/ntr/ntq051. PMID 20889477
- [Background] Smit ES, Fidler JA, West R. The role of desire, duty and intention in predicting attempts to quit smoking. Addiction. 2011 Apr;106(4):844-51. doi: 10.1111/j.1360-0443.2010.03317.x. Epub 2011 Feb 14. PMID 21205048
- [Background] Albano JD, Ward E, Jemal A, Anderson R, Cokkinides VE, Murray T, Henley J, Liff J, Thun MJ. Cancer mortality in the United States by education level and race. J Natl Cancer Inst. 2007 Sep 19;99(18):1384-94. doi: 10.1093/jnci/djm127. Epub 2007 Sep 11. PMID 17848670
- [Background] Siahpush M. Socioeconomic status and tobacco expenditure among Australian households: results from the 1998-99 Household Expenditure Survey. J Epidemiol Community Health. 2003 Oct;57(10):798-801. doi: 10.1136/jech.57.10.798. PMID 14573585
- [Background] Shelley D, Cantrell MJ, Moon-Howard J, Ramjohn DQ, VanDevanter N. The $5 man: the underground economic response to a large cigarette tax increase in New York City. Am J Public Health. 2007 Aug;97(8):1483-8. doi: 10.2105/AJPH.2005.079921. Epub 2007 Jun 28. PMID 17600270
- [Background] Stead M, MacAskill S, MacKintosh AM, Reece J, Eadie D. "It's as if you're locked in": qualitative explanations for area effects on smoking in disadvantaged communities. Health Place. 2001 Dec;7(4):333-43. doi: 10.1016/s1353-8292(01)00025-9. PMID 11682332
- [Background] Siahpush M, Borland R, Scollo M. Smoking and financial stress. Tob Control. 2003 Mar;12(1):60-6. doi: 10.1136/tc.12.1.60. PMID 12612364
- [Background] Semba RD, Kalm LM, de Pee S, Ricks MO, Sari M, Bloem MW. Paternal smoking is associated with increased risk of child malnutrition among poor urban families in Indonesia. Public Health Nutr. 2007 Jan;10(1):7-15. doi: 10.1017/S136898000722292X. PMID 17212837
- [Background] Cutler-Triggs C, Fryer GE, Miyoshi TJ, Weitzman M. Increased rates and severity of child and adult food insecurity in households with adult smokers. Arch Pediatr Adolesc Med. 2008 Nov;162(11):1056-62. doi: 10.1001/archpediatrics.2008.2. PMID 18981354
- [Background] Chaloupka FJ. Smoking, food insecurity, and tobacco control. Arch Pediatr Adolesc Med. 2008 Nov;162(11):1096-8. doi: 10.1001/archpedi.162.11.1096. No abstract available. PMID 18981362
- [Background] Carpenter MJ, Ford ME, Cartmell K, Alberg AJ. Misperceptions of nicotine replacement therapy within racially and ethnically diverse smokers. J Natl Med Assoc. 2011 Sep-Oct;103(9-10):885-94. doi: 10.1016/s0027-9684(15)30444-2. PMID 22364057
- [Background] McAfee TA. Quitlines a tool for research and dissemination of evidence-based cessation practices. Am J Prev Med. 2007 Dec;33(6 Suppl):S357-67. doi: 10.1016/j.amepre.2007.09.011. PMID 18021911
- [Background] Cummins SE, Bailey L, Campbell S, Koon-Kirby C, Zhu SH. Tobacco cessation quitlines in North America: a descriptive study. Tob Control. 2007 Dec;16 Suppl 1(Suppl 1):i9-15. doi: 10.1136/tc.2007.020370. PMID 18048639
- [Background] Zhu SH, Anderson CM, Tedeschi GJ, Rosbrook B, Johnson CE, Byrd M, Gutierrez-Terrell E. Evidence of real-world effectiveness of a telephone quitline for smokers. N Engl J Med. 2002 Oct 3;347(14):1087-93. doi: 10.1056/NEJMsa020660. PMID 12362011
- [Background] Cummings KM, Hyland A, Fix B, Bauer U, Celestino P, Carlin-Menter S, Miller N, Frieden TR. Free nicotine patch giveaway program 12-month follow-up of participants. Am J Prev Med. 2006 Aug;31(2):181-4. doi: 10.1016/j.amepre.2006.03.027. Epub 2006 Jun 12. PMID 16829336
- [Background] Cummings KM, Fix B, Celestino P, Carlin-Menter S, O'Connor R, Hyland A. Reach, efficacy, and cost-effectiveness of free nicotine medication giveaway programs. J Public Health Manag Pract. 2006 Jan-Feb;12(1):37-43. doi: 10.1097/00124784-200601000-00009. PMID 16340514
- [Background] Bauer JE, Carlin-Menter SM, Celestino PB, Hyland A, Cummings KM. Giving away free nicotine medications and a cigarette substitute (Better Quit) to promote calls to a quitline. J Public Health Manag Pract. 2006 Jan-Feb;12(1):60-7. doi: 10.1097/00124784-200601000-00012. PMID 16340517
- [Background] Ross JS, Bradley EH, Busch SH. Use of health care services by lower-income and higher-income uninsured adults. JAMA. 2006 May 3;295(17):2027-36. doi: 10.1001/jama.295.17.2027. PMID 16670411
- [Background] Ross JS, Bernheim SM, Bradley EH, Teng HM, Gallo WT. Use of preventive care by the working poor in the United States. Prev Med. 2007 Mar;44(3):254-9. doi: 10.1016/j.ypmed.2006.11.006. Epub 2006 Dec 29. PMID 17196642
- [Background] Kerner JF, Dusenbury L, Mandelblatt JS. Poverty and cultural diversity: challenges for health promotion among the medically underserved. Annu Rev Public Health. 1993;14:355-77. doi: 10.1146/annurev.pu.14.050193.002035. No abstract available. PMID 8323594
- [Background] Chisholm JS, Burbank VK. Evolution and inequality. Int J Epidemiol. 2001 Apr;30(2):206-11. doi: 10.1093/ije/30.2.206. PMID 11369714
- [Background] Zhang L, Vickerman K, Malarcher A, Carpenter K. Changes in Quitline Caller Characteristics During a National Tobacco Education Campaign. Nicotine Tob Res. 2015 Sep;17(9):1161-6. doi: 10.1093/ntr/ntu271. Epub 2015 Jan 5. PMID 25561612
- [Background] Duke JC, Mann N, Davis KC, MacMonegle A, Allen J, Porter L. The impact of a state-sponsored mass media campaign on use of telephone quitline and web-based cessation services. Prev Chronic Dis. 2014 Dec 24;11:E225. doi: 10.5888/pcd11.140354. PMID 25539129
- [Background] Arkin EB, Romano RM, Van Nevel JP, McKenna JW. Effect of the mass media in promoting calls to the Cancer Information Service. J Natl Cancer Inst Monogr. 1993;(14):35-43. PMID 8123357
- [Background] Boyd NR, Sutton C, Orleans CT, McClatchey MW, Bingler R, Fleisher L, Heller D, Baum S, Graves C, Ward JA. Quit Today! A targeted communications campaign to increase use of the cancer information service by African American smokers. Prev Med. 1998 Sep-Oct;27(5 Pt 2):S50-60. doi: 10.1006/pmed.1998.0383. PMID 9808824
- [Background] Centers for Disease Control and Prevention (CDC). Impact of a national tobacco education campaign on weekly numbers of quitline calls and website visitors--United States, March 4-June 23, 2013. MMWR Morb Mortal Wkly Rep. 2013 Sep 20;62(37):763-7. PMID 24048152
- [Background] Niederdeppe J, Kuang X, Crock B, Skelton A. Media campaigns to promote smoking cessation among socioeconomically disadvantaged populations: what do we know, what do we need to learn, and what should we do now? Soc Sci Med. 2008 Nov;67(9):1343-55. doi: 10.1016/j.socscimed.2008.06.037. Epub 2008 Aug 7. PMID 18691793
- [Background] Yano EM, Rubenstein LV, Farmer MM, Chernof BA, Mittman BS, Lanto AB, Simon BF, Lee ML, Sherman SE. Targeting primary care referrals to smoking cessation clinics does not improve quit rates: implementing evidence-based interventions into practice. Health Serv Res. 2008 Oct;43(5 Pt 1):1637-61. doi: 10.1111/j.1475-6773.2008.00865.x. Epub 2008 Jun 3. PMID 18522670
- [Background] Sherman SE, Joseph AM, Yano EM, Simon BF, Arikian N, Rubenstein LV, Parkerton P, Mittman BS. Assessing the institutional approach to implementing smoking cessation practice guidelines in veterans health administration facilities. Mil Med. 2006 Jan;171(1):80-7. doi: 10.7205/milmed.171.1.80. PMID 16532880
- [Background] Ward MM, Doebbeling BN, Vaughn TE, Uden-Holman T, Clarke WR, Woolson RF, Letuchy E, Branch LG, Perlin J. Effectiveness of a nationally implemented smoking cessation guideline on provider and patient practices. Prev Med. 2003 Mar;36(3):265-71. doi: 10.1016/s0091-7435(02)00046-4. PMID 12634017
- [Background] Sorensen G, Stoddard A, Ockene JK, Hunt MK, Youngstrom R. Worker participation in an integrated health promotion/health protection program: results from the WellWorks project. Health Educ Q. 1996 May;23(2):191-203. doi: 10.1177/109019819602300205. PMID 8744872
- [Background] Walsh DC, Jennings SE, Mangione T, Merrigan DM. Health promotion versus health protection? Employees' perceptions and concerns. J Public Health Policy. 1991 Summer;12(2):148-64. PMID 1885757
- [Background] Green KL. Issues of control and responsibility in workers' health. Health Educ Q. 1988 Winter;15(4):473-86. doi: 10.1177/109019818801500407. PMID 3230020
- [Background] Senn TE, Walsh JL, Carey MP. The mediating roles of perceived stress and health behaviors in the relation between objective, subjective, and neighborhood socioeconomic status and perceived health. Ann Behav Med. 2014 Oct;48(2):215-24. doi: 10.1007/s12160-014-9591-1. PMID 24648016
- [Background] Remler DK, Glied SA. What other programs can teach us: increasing participation in health insurance programs. Am J Public Health. 2003 Jan;93(1):67-74. doi: 10.2105/ajph.93.1.67. PMID 12511389
- [Background] Beaglehole R. International trends in coronary heart disease mortality, morbidity, and risk factors. Epidemiol Rev. 1990;12:1-15. doi: 10.1093/oxfordjournals.epirev.a036048. No abstract available. PMID 2286214
- [Background] Link BG, Phelan J. Social conditions as fundamental causes of disease. J Health Soc Behav. 1995;Spec No:80-94. PMID 7560851
- [Background] Melchior M, Caspi A, Howard LM, Ambler AP, Bolton H, Mountain N, Moffitt TE. Mental health context of food insecurity: a representative cohort of families with young children. Pediatrics. 2009 Oct;124(4):e564-72. doi: 10.1542/peds.2009-0583. Epub 2009 Sep 28. PMID 19786424
- [Background] Blazer DG, Sachs-Ericsson N, Hybels CF. Perception of unmet basic needs as a predictor of depressive symptoms among community-dwelling older adults. J Gerontol A Biol Sci Med Sci. 2007 Feb;62(2):191-5. doi: 10.1093/gerona/62.2.191. PMID 17339645
- [Background] Sachs-Ericsson N, Schatschneider C, Blazer DG. Perception of unmet basic needs as a predictor of physical functioning among community-dwelling older adults. J Aging Health. 2006 Dec;18(6):852-68. doi: 10.1177/0898264306293261. PMID 17099137
- [Background] Blazer DG, Sachs-Ericsson N, Hybels CF. Perception of unmet basic needs as a predictor of mortality among community-dwelling older adults. Am J Public Health. 2005 Feb;95(2):299-304. doi: 10.2105/AJPH.2003.035576. PMID 15671468
- [Background] Taylor SE, Repetti RL, Seeman T. Health psychology: what is an unhealthy environment and how does it get under the skin? Annu Rev Psychol. 1997;48:411-47. doi: 10.1146/annurev.psych.48.1.411. PMID 9046565
- [Background] Lynch JW, Kaplan GA, Shema SJ. Cumulative impact of sustained economic hardship on physical, cognitive, psychological, and social functioning. N Engl J Med. 1997 Dec 25;337(26):1889-95. doi: 10.1056/NEJM199712253372606. PMID 9407157
- [Background] Kushel MB, Gupta R, Gee L, Haas JS. Housing instability and food insecurity as barriers to health care among low-income Americans. J Gen Intern Med. 2006 Jan;21(1):71-7. doi: 10.1111/j.1525-1497.2005.00278.x. PMID 16423128
- [Background] Timmerman GM, Acton GJ. The relationship between basic need satisfaction and emotional eating. Issues Ment Health Nurs. 2001 Oct-Nov;22(7):691-701. doi: 10.1080/016128401750434482. PMID 11881182
- [Background] Acton GJ, Malathum P. Basic need status and health-promoting self-care behavior in adults. West J Nurs Res. 2000 Nov;22(7):796-811. doi: 10.1177/01939450022044764. PMID 11077548
- [Background] Fitzpatrick-Lewis D, Ganann R, Krishnaratne S, Ciliska D, Kouyoumdjian F, Hwang SW. Effectiveness of interventions to improve the health and housing status of homeless people: a rapid systematic review. BMC Public Health. 2011 Aug 10;11:638. doi: 10.1186/1471-2458-11-638. PMID 21831318
- [Background] Wolitski RJ, Kidder DP, Pals SL, Royal S, Aidala A, Stall R, Holtgrave DR, Harre D, Courtenay-Quirk C; Housing and Health Study Team. Randomized trial of the effects of housing assistance on the health and risk behaviors of homeless and unstably housed people living with HIV. AIDS Behav. 2010 Jun;14(3):493-503. doi: 10.1007/s10461-009-9643-x. PMID 19949848
- [Background] Thomson H, Thomas S, Sellstrom E, Petticrew M. The health impacts of housing improvement: a systematic review of intervention studies from 1887 to 2007. Am J Public Health. 2009 Nov;99 Suppl 3(Suppl 3):S681-92. doi: 10.2105/AJPH.2008.143909. PMID 19890174
- [Background] Leventhal T, Brooks-Gunn J. Moving to opportunity: an experimental study of neighborhood effects on mental health. Am J Public Health. 2003 Sep;93(9):1576-82. doi: 10.2105/ajph.93.9.1576. PMID 12948983
- [Background] Williams DR, Costa MV, Odunlami AO, Mohammed SA. Moving upstream: how interventions that address the social determinants of health can improve health and reduce disparities. J Public Health Manag Pract. 2008 Nov;14 Suppl(Suppl):S8-17. doi: 10.1097/01.PHH.0000338382.36695.42. PMID 18843244
- [Background] Weinstein ND, Marcus SE, Moser RP. Smokers' unrealistic optimism about their risk. Tob Control. 2005 Feb;14(1):55-9. doi: 10.1136/tc.2004.008375. PMID 15735301
- [Background] Smedley BD, Syme SL; Committee on Capitalizing on Social Science and Behavioral Research to Improve the Public's Health. Promoting health: intervention strategies from social and behavioral research. Am J Health Promot. 2001 Jan-Feb;15(3):149-66. doi: 10.4278/0890-1171-15.3.149. PMID 11265579
- [Background] Wylie-Rosett J, Herman WH, Goldberg RB. Lifestyle intervention to prevent diabetes: intensive and cost effective. Curr Opin Lipidol. 2006 Feb;17(1):37-44. doi: 10.1097/01.mol.0000203890.27267.eb. PMID 16407714
- [Background] Drewnowski A, Darmon N. The economics of obesity: dietary energy density and energy cost. Am J Clin Nutr. 2005 Jul;82(1 Suppl):265S-273S. doi: 10.1093/ajcn/82.1.265S. PMID 16002835
- [Background] Herman WH, Hoerger TJ, Brandle M, Hicks K, Sorensen S, Zhang P, Hamman RF, Ackermann RT, Engelgau MM, Ratner RE; Diabetes Prevention Program Research Group. The cost-effectiveness of lifestyle modification or metformin in preventing type 2 diabetes in adults with impaired glucose tolerance. Ann Intern Med. 2005 Mar 1;142(5):323-32. doi: 10.7326/0003-4819-142-5-200503010-00007. PMID 15738451
- [Background] Klesges LM, Dzewaltowski DA, Glasgow RE. Review of external validity reporting in childhood obesity prevention research. Am J Prev Med. 2008 Mar;34(3):216-23. doi: 10.1016/j.amepre.2007.11.019. PMID 18312810
- [Background] Glasgow RE, Green LW, Klesges LM, Abrams DB, Fisher EB, Goldstein MG, Hayman LL, Ockene JK, Orleans CT. External validity: we need to do more. Ann Behav Med. 2006 Apr;31(2):105-8. doi: 10.1207/s15324796abm3102_1. No abstract available. PMID 16542124
- [Background] Glasgow RE, Klesges LM, Dzewaltowski DA, Estabrooks PA, Vogt TM. Evaluating the impact of health promotion programs: using the RE-AIM framework to form summary measures for decision making involving complex issues. Health Educ Res. 2006 Oct;21(5):688-94. doi: 10.1093/her/cyl081. Epub 2006 Aug 31. PMID 16945984
- [Background] Gusi N, Reyes MC, Gonzalez-Guerrero JL, Herrera E, Garcia JM. Cost-utility of a walking programme for moderately depressed, obese, or overweight elderly women in primary care: a randomised controlled trial. BMC Public Health. 2008 Jul 8;8:231. doi: 10.1186/1471-2458-8-231. PMID 18611277
- [Background] Urbanski P, Wolf A, Herman WH. Cost-effectiveness of diabetes education. J Am Diet Assoc. 2008 Apr;108(4 Suppl 1):S6-11. doi: 10.1016/j.jada.2008.01.019. PMID 18358259
- [Background] Windyga P, Kim K, White V, Leon M, Bag A, Chen W. Cost-return prediction in morbidly obese employees following weight loss interventions: a study framework. Annu Int Conf IEEE Eng Med Biol Soc. 2007;2007:1766-9. doi: 10.1109/IEMBS.2007.4352653. PMID 18002319
- [Background] Brown HS 3rd, Perez A, Li YP, Hoelscher DM, Kelder SH, Rivera R. The cost-effectiveness of a school-based overweight program. Int J Behav Nutr Phys Act. 2007 Oct 1;4:47. doi: 10.1186/1479-5868-4-47. PMID 17908315
- [Background] Kreuter MW. Reach, effectiveness, and connections: the case for partnering with 2-1-1 to eliminate health disparities. Am J Prev Med. 2012 Dec;43(6 Suppl 5):S420-1. doi: 10.1016/j.amepre.2012.09.024. No abstract available. PMID 23157759
- [Background] McQueen A, Kreuter MW. Women's cognitive and affective reactions to breast cancer survivor stories: a structural equation analysis. Patient Educ Couns. 2010 Dec;81 Suppl:S15-21. doi: 10.1016/j.pec.2010.08.015. Epub 2010 Sep 17. PMID 20850258
- [Background] McQueen A, Kreuter MW, Kalesan B, Alcaraz KI. Understanding narrative effects: the impact of breast cancer survivor stories on message processing, attitudes, and beliefs among African American women. Health Psychol. 2011 Nov;30(6):674-82. doi: 10.1037/a0025395. Epub 2011 Sep 5. PMID 21895370
- [Background] McQueen A, Swank PR, Bastian LA, Vernon SW. Predictors of perceived susceptibility of breast cancer and changes over time: a mixed modeling approach. Health Psychol. 2008 Jan;27(1):68-77. doi: 10.1037/0278-6133.27.1.68. PMID 18230016
- [Background] McQueen A, Vernon SW, Myers RE, Watts BG, Lee ES, Tilley BC. Correlates and predictors of colorectal cancer screening among male automotive workers. Cancer Epidemiol Biomarkers Prev. 2007 Mar;16(3):500-9. doi: 10.1158/1055-9965.EPI-06-0757. PMID 17372245
- [Background] McQueen A, Tiro JA, Vernon SW. Construct validity and invariance of four factors associated with colorectal cancer screening across gender, race, and prior screening. Cancer Epidemiol Biomarkers Prev. 2008 Sep;17(9):2231-7. doi: 10.1158/1055-9965.EPI-08-0176. PMID 18768488
- [Background] McQueen A, Vernon SW, Rothman AJ, Norman GJ, Myers RE, Tilley BC. Examining the role of perceived susceptibility on colorectal cancer screening intention and behavior. Ann Behav Med. 2010 Oct;40(2):205-17. doi: 10.1007/s12160-010-9215-3. PMID 20658212
- [Background] McQueen A, Vernon SW, Swank PR. Construct definition and scale development for defensive information processing: an application to colorectal cancer screening. Health Psychol. 2013 Feb;32(2):190-202. doi: 10.1037/a0027311. Epub 2012 Feb 20. PMID 22353026
- [Background] McQueen A, Tower S, Sumner W. Interviews with "vapers": implications for future research with electronic cigarettes. Nicotine Tob Res. 2011 Sep;13(9):860-7. doi: 10.1093/ntr/ntr088. Epub 2011 May 12. PMID 21571692
- [Background] McQueen A, Bartholomew LK, Greisinger AJ, Medina GG, Hawley ST, Haidet P, Bettencourt JL, Shokar NK, Ling BS, Vernon SW. Behind closed doors: physician-patient discussions about colorectal cancer screening. J Gen Intern Med. 2009 Nov;24(11):1228-35. doi: 10.1007/s11606-009-1108-4. Epub 2009 Sep 18. PMID 19763699
- [Background] Medina GG, McQueen A, Greisinger AJ, Bartholomew LK, Vernon SW. What would make getting colorectal cancer screening easier? Perspectives from screeners and nonscreeners. Gastroenterol Res Pract. 2012;2012:895807. doi: 10.1155/2012/895807. Epub 2012 Jan 4. PMID 22272194
- [Background] McQueen A, Kreuter MW, Boyum S, Thompson VS, Caburnay CA, Waters EA, Kaphingst KA, Rath S, Fu Q. Reactions to FDA-Proposed Graphic Warning Labels Affixed to U.S. Smokers' Cigarette Packs. Nicotine Tob Res. 2015 Jul;17(7):784-95. doi: 10.1093/ntr/ntu339. Epub 2015 Jan 14. PMID 25589676
- [Background] Kreuter MW, Caburnay CA, Chen JJ, Donlin MJ. Effectiveness of individually tailored calendars in promoting childhood immunization in urban public health centers. Am J Public Health. 2004 Jan;94(1):122-7. doi: 10.2105/ajph.94.1.122. PMID 14713709
- [Background] Caburnay CA, Kreuter MW, Cameron G, Luke DA, Cohen EL, McDaniels L, Wohlberg M, Atkins P. Black newspapers as a tool for cancer education in African American communities. Ethn Dis. 2008 Autumn;18(4):488-95. PMID 19157255
- [Background] Caburnay CA, Luke DA, Cameron GT, Cohen EL, Fu Q, Lai CL, Stemmle JT, Paulen M, Jackson L, Kreuter MW. Evaluating the Ozioma cancer news service: a community randomized trial in 24 U.S. cities. Prev Med. 2012 Jun;54(6):425-30. doi: 10.1016/j.ypmed.2012.04.010. Epub 2012 Apr 23. PMID 22546317
- [Background] Fellows JL, Bush T, McAfee T, Dickerson J. Cost effectiveness of the Oregon quitline "free patch initiative". Tob Control. 2007 Dec;16 Suppl 1(Suppl 1):i47-52. doi: 10.1136/tc.2007.019943. PMID 18048632
- [Background] Alcaraz KI, Arnold LD, Eddens KS, Lai C, Rath S, Greer R, Kreuter MW. Exploring 2-1-1 service requests as potential markers for cancer control needs. Am J Prev Med. 2012 Dec;43(6 Suppl 5):S469-74. doi: 10.1016/j.amepre.2012.08.019. PMID 23157767
- [Background] Eddens KS, Alcaraz KI, Kreuter MW, Rath S, Greer R. A 2-1-1 research collaboration: participant accrual and service quality indicators. Am J Prev Med. 2012 Dec;43(6 Suppl 5):S483-9. doi: 10.1016/j.amepre.2012.09.007. PMID 23157769
- [Background] Wiehagen T, Caito NM, Thompson VS, Casey CM, Weaver NL, Jupka K, Kreuter MW. Applying projective techniques to formative research in health communication development. Health Promot Pract. 2007 Apr;8(2):164-72. doi: 10.1177/1524839906289818. Epub 2006 Sep 26. PMID 17003247
- [Background] Boslaugh SE, Kreuter MW, Nicholson RA, Naleid K. Comparing demographic, health status and psychosocial strategies of audience segmentation to promote physical activity. Health Educ Res. 2005 Aug;20(4):430-8. doi: 10.1093/her/cyg138. Epub 2004 Nov 30. PMID 15572439
- [Background] Nicholson RA, Kreuter MW, Lapka C, Wellborn R, Clark EM, Sanders-Thompson V, Jacobsen HM, Casey C. Unintended effects of emphasizing disparities in cancer communication to African-Americans. Cancer Epidemiol Biomarkers Prev. 2008 Nov;17(11):2946-53. doi: 10.1158/1055-9965.EPI-08-0101. PMID 18990735
- [Background] Sanders Thompson VL, Cavazos-Rehg PA, Jupka K, Caito N, Gratzke J, Tate KY, Deshpande A, Kreuter MW. Evidential preferences: cultural appropriateness strategies in health communications. Health Educ Res. 2008 Jun;23(3):549-59. doi: 10.1093/her/cym029. Epub 2007 Jul 13. PMID 17631608
- [Background] Kreuter MW, Wray RJ. Tailored and targeted health communication: strategies for enhancing information relevance. Am J Health Behav. 2003 Nov-Dec;27 Suppl 3:S227-32. doi: 10.5993/ajhb.27.1.s3.6. PMID 14672383
- [Background] Kreuter MW, Black WJ, Friend L, Booker AC, Klump P, Bobra S, Holt CL. Use of computer kiosks for breast cancer education in five community settings. Health Educ Behav. 2006 Oct;33(5):625-42. doi: 10.1177/1090198106290795. Epub 2006 Aug 21. PMID 16923835
- [Background] Kreuter MW, Sugg-Skinner C, Holt CL, Clark EM, Haire-Joshu D, Fu Q, Booker AC, Steger-May K, Bucholtz D. Cultural tailoring for mammography and fruit and vegetable intake among low-income African-American women in urban public health centers. Prev Med. 2005 Jul;41(1):53-62. doi: 10.1016/j.ypmed.2004.10.013. Epub 2004 Nov 26. PMID 15916993
- [Background] Kreuter MW, Skinner CS, Steger-May K, Holt CL, Bucholtz DC, Clark EM, Haire-Joshu D. Responses to behaviorally vs culturally tailored cancer communication among African American women. Am J Health Behav. 2004 May-Jun;28(3):195-207. doi: 10.5993/ajhb.28.3.1. PMID 15152880
- [Background] Kreuter MW, Steger-May K, Bobra S, Booker A, Holt CL, Lukwago SN, Skinner CS. Sociocultural characteristics and responses to cancer education materials among African American women. Cancer Control. 2003 Sep-Oct;10(5 Suppl):69-80. doi: 10.1177/107327480301005s10. PMID 14581907
- [Background] Eddens KS, Kreuter MW. Proactive screening for health needs in United Way's 2-1-1 information and referral service. J Soc Serv Res. 2011;37(2):113-123. doi: 10.1080/01488376.2011.547445. PMID 21566702
- [Background] Kreuter MW, Alcaraz KI, Pfeiffer D, Christopher K. Using dissemination research to identify optimal community settings for tailored breast cancer information kiosks. J Public Health Manag Pract. 2008 Mar-Apr;14(2):160-9. doi: 10.1097/01.PHH.0000311895.57831.02. PMID 18287923
- [Background] Kreuter MW, Lukwago SN, Bucholtz RD, Clark EM, Sanders-Thompson V. Achieving cultural appropriateness in health promotion programs: targeted and tailored approaches. Health Educ Behav. 2003 Apr;30(2):133-46. doi: 10.1177/1090198102251021. PMID 12693519
- [Background] Kreuter MW, McClure SM. The role of culture in health communication. Annu Rev Public Health. 2004;25:439-55. doi: 10.1146/annurev.publhealth.25.101802.123000. PMID 15015929
- [Background] Deshpande AD, Sanders Thompson VL, Vaughn KP, Kreuter MW. The use of sociocultural constructs in cancer screening research among African Americans. Cancer Control. 2009 Jul;16(3):256-65. doi: 10.1177/107327480901600308. PMID 19556966
- [Background] Strecher VJ, Kreuter M, Den Boer DJ, Kobrin S, Hospers HJ, Skinner CS. The effects of computer-tailored smoking cessation messages in family practice settings. J Fam Pract. 1994 Sep;39(3):262-70. PMID 8077905
- [Background] McQueen A, Shacham E, Sumner W, Overton ET. Beliefs, experience, and interest in pharmacotherapy among smokers with HIV. Am J Health Behav. 2014 Mar;38(2):284-96. doi: 10.5993/AJHB.38.2.14. PMID 24629557
- [Background] Linnan LA. Research collaboration with 2-1-1 to eliminate health disparities: an introduction. Am J Prev Med. 2012 Dec;43(6 Suppl 5):S415-9. doi: 10.1016/j.amepre.2012.09.025. No abstract available. PMID 23157758
- [Background] Kegler MC, Bundy L, Haardorfer R, Escoffery C, Berg C, Yembra D, Kreuter M, Hovell M, Williams R, Mullen PD, Ribisl K, Burnham D. A minimal intervention to promote smoke-free homes among 2-1-1 callers: a randomized controlled trial. Am J Public Health. 2015 Mar;105(3):530-7. doi: 10.2105/AJPH.2014.302260. Epub 2015 Jan 20. PMID 25602863
- [Background] Purnell JQ, Kreuter MW, Eddens KS, Ribisl KM, Hannon P, Williams RS, Fernandez ME, Jobe D, Gemmel S, Morris M, Fagin D. Cancer control needs of 2-1-1 callers in Missouri, North Carolina, Texas, and Washington. J Health Care Poor Underserved. 2012 May;23(2):752-67. doi: 10.1353/hpu.2012.0061. PMID 22643622
- [Background] Daily LS. Health research and surveillance potential to partner with 2-1-1. Am J Prev Med. 2012 Dec;43(6 Suppl 5):S422-4. doi: 10.1016/j.amepre.2012.09.021. No abstract available. PMID 23157760
- [Background] Rodgers JT, Purnell JQ. Healthcare navigation service in 2-1-1 San Diego: guiding individuals to the care they need. Am J Prev Med. 2012 Dec;43(6 Suppl 5):S450-6. doi: 10.1016/j.amepre.2012.08.012. PMID 23157764
- [Background] Roux AM, Herrera P, Wold CM, Dunkle MC, Glascoe FP, Shattuck PT. Developmental and autism screening through 2-1-1: reaching underserved families. Am J Prev Med. 2012 Dec;43(6 Suppl 5):S457-63. doi: 10.1016/j.amepre.2012.08.011. PMID 23157765
- [Background] Cortinois AA, Glazier RH, Caidi N, Andrews G, Herbert-Copley M, Jadad AR. Toronto's 2-1-1 healthcare services for immigrant populations. Am J Prev Med. 2012 Dec;43(6 Suppl 5):S475-82. doi: 10.1016/j.amepre.2012.08.010. PMID 23157768
- [Background] Savas LS, Fernandez ME, Jobe D, Carmack CC. Human papillomavirus vaccine: 2-1-1 helplines and minority parent decision-making. Am J Prev Med. 2012 Dec;43(6 Suppl 5):S490-6. doi: 10.1016/j.amepre.2012.09.003. PMID 23157770
- [Background] Finney Rutten LJ, Augustson EM, Moser RP, Beckjord EB, Hesse BW. Smoking knowledge and behavior in the United States: sociodemographic, smoking status, and geographic patterns. Nicotine Tob Res. 2008 Oct;10(10):1559-70. doi: 10.1080/14622200802325873. PMID 18946775
- [Background] Wogalter MS, Conzola VC, Smith-Jackson TL. Research-based guidelines for warning design and evaluation. Appl Ergon. 2002 May;33(3):219-30. doi: 10.1016/s0003-6870(02)00009-1. PMID 12164506
- [Background] Deprey M, McAfee T, Bush T, McClure JB, Zbikowski S, Mahoney L. Using free patches to improve reach of the Oregon Quit Line. J Public Health Manag Pract. 2009 Sep-Oct;15(5):401-8. doi: 10.1097/PHH.0b013e3181952345. PMID 19704308
- [Background] Bush T, Levine MD, Zbikowski S, Deprey M, Rabius V, McAfee T, Wiatrek DE. Weight Gain After Quitting: Attitudes, Beliefs and Counselling Strategies of Cessation Counsellors. J Smok Cessat. 2008 Dec;3(2):124-132. doi: 10.1375/jsc.3.2.124. PMID 20574550
- [Background] Morris N, Gilpin DR, Lenos M, Hobbs R. Interpretations of cigarette advertisement warning labels by Philadelphia Puerto Ricans. J Health Commun. 2011 Sep;16(8):908-22. doi: 10.1080/10810730.2011.561910. Epub 2011 May 24. PMID 21534024
- [Background] Wakefield M, Bayly M, Durkin S, Cotter T, Mullin S, Warne C; International Anti-Tobacco Advertisement Rating Study Team. Smokers' responses to television advertisements about the serious harms of tobacco use: pre-testing results from 10 low- to middle-income countries. Tob Control. 2013 Jan;22(1):24-31. doi: 10.1136/tobaccocontrol-2011-050171. Epub 2011 Oct 12. PMID 21994276
- [Background] McCool J, Webb L, Cameron LD, Hoek J. Graphic warning labels on plain cigarette packs: will they make a difference to adolescents? Soc Sci Med. 2012 Apr;74(8):1269-73. doi: 10.1016/j.socscimed.2011.12.043. Epub 2012 Feb 17. PMID 22385817
- [Background] Mutti S, Hammond D, Reid JL, Thrasher JF. The efficacy of cigarette warning labels on health beliefs in the United States and Mexico. J Health Commun. 2013;18(10):1180-92. doi: 10.1080/10810730.2013.778368. Epub 2013 Aug 1. PMID 23905611
- [Background] Hammond D, Fong GT, McNeill A, Borland R, Cummings KM. Effectiveness of cigarette warning labels in informing smokers about the risks of smoking: findings from the International Tobacco Control (ITC) Four Country Survey. Tob Control. 2006 Jun;15 Suppl 3(Suppl 3):iii19-25. doi: 10.1136/tc.2005.012294. PMID 16754942
- [Background] Magnan RE, Cameron LD. Do Young Adults Perceive That Cigarette Graphic Warnings Provide New Knowledge About the Harms of Smoking? Ann Behav Med. 2015 Aug;49(4):594-604. doi: 10.1007/s12160-015-9691-6. PMID 25697134
- [Background] Sussenbach P, Niemeier S, Glock S. Effects of and attention to graphic warning labels on cigarette packages. Psychol Health. 2013;28(10):1192-206. doi: 10.1080/08870446.2013.799161. Epub 2013 May 29. PMID 23713958
- [Background] Curry SJ, Grothaus L, McBride C. Reasons for quitting: intrinsic and extrinsic motivation for smoking cessation in a population-based sample of smokers. Addict Behav. 1997 Nov-Dec;22(6):727-39. doi: 10.1016/s0306-4603(97)00059-2. PMID 9426790
- [Background] McCaul KD, Hockemeyer JR, Johnson RJ, Zetocha K, Quinlan K, Glasgow RE. Motivation to quit using cigarettes: a review. Addict Behav. 2006 Jan;31(1):42-56. doi: 10.1016/j.addbeh.2005.04.004. PMID 15916861
- [Background] Gwaltney CJ, Metrik J, Kahler CW, Shiffman S. Self-efficacy and smoking cessation: a meta-analysis. Psychol Addict Behav. 2009 Mar;23(1):56-66. doi: 10.1037/a0013529. PMID 19290690
- [Background] Javitz HS, Zbikowski SM, Deprey M, McAfee TA, McClure JB, Richards J, Catz SL, Jack LM, Swan GE. Cost-effectiveness of varenicline and three different behavioral treatment formats for smoking cessation. Transl Behav Med. 2011 Mar 1;1(1):182-190. doi: 10.1007/s13142-010-0009-8. PMID 21731592
- [Background] Javitz HS, Swan GE, Zbikowski SM, Curry SJ, McAfee TA, Decker DL, Patterson R, Jack LM. Cost-effectiveness of different combinations of bupropion SR dose and behavioral treatment for smoking cessation: a societal perspective. Am J Manag Care. 2004 Mar;10(3):217-26. PMID 15032259
- [Background] Javitz HS, Swan GE, Zbikowski SM, Curry SJ, McAfee TA, Decker D, Patterson R, Jack LM. Return on investment of different combinations of bupropion SR dose and behavioral treatment for smoking cessation in a health care setting: an employer's perspective. Value Health. 2004 Sep-Oct;7(5):535-43. doi: 10.1111/j.1524-4733.2004.75005.x. PMID 15367249
- [Background] Campbell HS, Ossip-Klein D, Bailey L, Saul J; North American Quitline Consortium. Minimal dataset for quitlines: a best practice. Tob Control. 2007 Dec;16 Suppl 1(Suppl 1):i16-20. doi: 10.1136/tc.2007.019976. PMID 18048624
- [Background] Shea S, Stein AD, Lantigua R, Basch CE. Reliability of the behavioral risk factor survey in a triethnic population. Am J Epidemiol. 1991 Mar 1;133(5):489-500. doi: 10.1093/oxfordjournals.aje.a115916. PMID 2000859
- [Background] Brownson RC, Eyler AA, King AC, Shyu YL, Brown DR, Homan SM. Reliability of information on physical activity and other chronic disease risk factors among US women aged 40 years or older. Am J Epidemiol. 1999 Feb 15;149(4):379-91. doi: 10.1093/oxfordjournals.aje.a009824. PMID 10025482
- [Background] Brownson RC, Jackson-Thompson J, Wilkerson JC, Kiani F. Reliability of information on chronic disease risk factors collected in the Missouri Behavioral Risk Factor Surveillance System. Epidemiology. 1994 Sep;5(5):545-9. PMID 7986871
- [Background] Nelson DE, Holtzman D, Bolen J, Stanwyck CA, Mack KA. Reliability and validity of measures from the Behavioral Risk Factor Surveillance System (BRFSS). Soz Praventivmed. 2001;46 Suppl 1:S3-42. PMID 11851091
- [Background] King AC, Cao D, Southard CC, Matthews A. Racial differences in eligibility and enrollment in a smoking cessation clinical trial. Health Psychol. 2011 Jan;30(1):40-8. doi: 10.1037/a0021649. PMID 21299293
- [Background] Cantrell J, Shelley D. Implementing a fax referral program for quitline smoking cessation services in urban health centers: a qualitative study. BMC Fam Pract. 2009 Dec 17;10:81. doi: 10.1186/1471-2296-10-81. PMID 20017930
- [Background] Weiss SM, Smith-Simone SY. Consumer and health literacy: The need to better design tobacco-cessation product packaging, labels, and inserts. Am J Prev Med. 2010 Mar;38(3 Suppl):S403-13. doi: 10.1016/j.amepre.2009.11.020. PMID 20176315
- [Background] Stevens AB, McDaniel KS, Glover ED, Wallace LS. Are instructions for over-the-counter nicotine replacement therapy products readable? Am J Health Behav. 2007 Sep-Oct;31 Suppl 1:S79-84. doi: 10.5555/ajhb.2007.31.supp.S79. PMID 17931140
- [Background] LESHAN LL. Time orientation and social class. J Abnorm Psychol. 1952 Jul;47(3):589-92. doi: 10.1037/h0056306. No abstract available. PMID 12980757
- [Background] Brown CM, Segal R. Ethnic differences in temporal orientation and its implications for hypertension management. J Health Soc Behav. 1996 Dec;37(4):350-61. PMID 8997890
- [Background] Rothspan S, Read SJ. Present versus future time perspective and HIV risk among heterosexual college students. Health Psychol. 1996 Mar;15(2):131-4. doi: 10.1037//0278-6133.15.2.131. PMID 8681921
- [Background] Lukwago SN, Kreuter MW, Holt CL, Steger-May K, Bucholtz DC, Skinner CS. Sociocultural correlates of breast cancer knowledge and screening in urban African American women. Am J Public Health. 2003 Aug;93(8):1271-4. doi: 10.2105/ajph.93.8.1271. No abstract available. PMID 12893610
- [Background] Smith KC, Stillman F, Bone L, Yancey N, Price E, Belin P, Kromm EE. Buying and selling "loosies" in Baltimore: the informal exchange of cigarettes in the community context. J Urban Health. 2007 Jul;84(4):494-507. doi: 10.1007/s11524-007-9189-z. PMID 17431795
- [Background] White VM, Gilpin EA, White MM, Pierce JP. How do smokers control their cigarette expenditures? Nicotine Tob Res. 2005 Aug;7(4):625-35. doi: 10.1080/14622200500184333. PMID 16085532
- [Background] Cavin SW, Pierce JP. Low-cost cigarettes and smoking behavior in California, 1990-1993. Am J Prev Med. 1996 Jan-Feb;12(1):17-21. PMID 8776290
- [Background] Klonoff EA, Fritz JM, Landrine H, Riddle RW, Tully-Payne L. The problem and sociocultural context of single-cigarette sales. JAMA. 1994 Feb 23;271(8):618-20. PMID 8301795
- [Background] Aloot CB, Vredevoe DL, Brecht ML. Evaluation of high-risk smoking practices used by the homeless. Cancer Nurs. 1993 Apr;16(2):123-30. PMID 8477400
- [Background] Centers for Disease Control and Prevention (CDC). Tobacco product use among middle and high school students--United States, 2011 and 2012. MMWR Morb Mortal Wkly Rep. 2013 Nov 15;62(45):893-7. PMID 24226625
- [Background] Sutherland C, Sullivan C, Bybee D. Effects of intimate partner violence versus poverty on women's health. Violence Against Women. 2001;7(10):1122-1143.
- [Background] Prochaska JO, Crimi P, Lapsanski D, Martel L, Reid P. Self-change processes, self-efficacy and self-concept in relapse and maintenance of cessation of smoking. Psychol Rep. 1982 Dec;51(3 Pt 1):983-90. doi: 10.2466/pr0.1982.51.3.983. No abstract available. PMID 7163454
- [Background] Velicer WF, DiClemente CC, Prochaska JO, Brandenburg N. Decisional balance measure for assessing and predicting smoking status. J Pers Soc Psychol. 1985 May;48(5):1279-89. doi: 10.1037//0022-3514.48.5.1279. PMID 3998990
- [Derived] Kreuter MW, Garg R, Fu Q, Caburnay C, Thompson T, Roberts C, Sandheinrich D, Javed I, Wolff JM, Butler T, Grimes LM, Carpenter KM, Pokojski R, Engelbrecht K, Howard V, McQueen A. Helping low-income smokers quit: findings from a randomized controlled trial comparing specialized quitline services with and without social needs navigation. Lancet Reg Health Am. 2023 Jun 24;23:100529. doi: 10.1016/j.lana.2023.100529. eCollection 2023 Jul. PMID 37408953
- [Derived] McQueen A, Wartts JG, Garg R, Carpenter KM, Kreuter MW. Leveling the Playing Field: Mailing Pharmacotherapy to Medicaid Members Who Smoke. Am J Prev Med. 2023 Feb;64(2):227-234. doi: 10.1016/j.amepre.2022.09.008. Epub 2022 Nov 3. PMID 36335079
- [Derived] Garg R, McQueen A, Roberts C, Butler T, Grimes LM, Thompson T, Caburnay C, Wolff J, Javed I, Carpenter KM, Wartts JG, Charles C, Howard V, Kreuter MW. Stress, depression, sleep problems and unmet social needs: Baseline characteristics of low-income smokers in a randomized cessation trial. Contemp Clin Trials Commun. 2021 Nov 11;24:100857. doi: 10.1016/j.conctc.2021.100857. eCollection 2021 Dec. PMID 34849423
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- Specialized Quitline With Basic Needs Navigator: Participants receive Specialized quitline services (see previous description) with navigator.
  Basic Needs Navigator: Navigators will: (1) identify and assess smokers' needs, including the reasons they called 2-1-1; (2) jointly generate solutions to address the needs; (3) develop plans to carry out the solutions, including; (4) help prioritize among multiple needs; (5) identify community resources that could help solve the problem; (6) determine eligibility for services; (7) help smokers access available resources by scheduling appointments and provide appointment reminders; (8) prepare smokers to interact with service agencies and/or act as an advocate on their behalf; (9) provide instrumental support such as arranging transportation; (10) actively intervene to resolve barriers to basic needs solutions; (11) oversee follow-up of problem solving actions; and (12) review progress made towards resolving unmet basic needs and adapt solutions accordingly.
Period: Overall Study
Arm/Group | Standard Quitline | Specialized Quitline | Standard Quitline With Basic Needs Navigator | Specialized Quitline With Basic Needs Navigator
Started | 485 | 485 | 484 | 490
Completed | 293 | 261 | 302 | 281
Not Completed | 192 | 224 | 182 | 209
Not completed — Death | 0 | 1 | 1 | 1
Not completed — Withdrawal by Subject | 24 | 27 | 7 | 22
Not completed — Lost to Follow-up | 168 | 196 | 174 | 186

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Quitline | Specialized Quitline | Standard Quitline With Basic Needs Navigator | Specialized Quitline With Basic Needs Navigator | Total
Number analyzed (Participants) | 485 | 485 | 484 | 490 | 1944
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.2 (12.1) | 49.0 (12.5) | 48.6 (12.2) | 47.8 (12.1) | 48.4 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 349 | 357 | 334 | 356 | 1396
  Male | 136 | 128 | 150 | 134 | 548
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 13 | 13 | 14 | 55
  Not Hispanic or Latino | 466 | 470 | 465 | 471 | 1872
  Unknown or Not Reported | 4 | 2 | 6 | 5 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 9 | 6 | 8 | 5 | 28
  Asian | 1 | 2 | 0 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1 | 2
  Black or African American | 268 | 278 | 275 | 290 | 1111
  White | 179 | 164 | 166 | 157 | 666
  More than one race | 25 | 29 | 25 | 28 | 107
  Unknown or Not Reported | 3 | 5 | 10 | 6 | 24

OUTCOME MEASURES:

1. Primary Outcome: Abstinence 6-months
Description: Report 7-day point prevalence abstinence measured at 6-months post --baseline
Time Frame: 6 months post-baseline
Population: Intention-to-treat sample
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Quitline | Specialized Quitline | Standard Quitline With Basic Needs Navigator | Specialized Quitline With Basic Needs Navigator
Number analyzed (Participants) | 485 | 485 | 484 | 490
Participants | 101 | 90 | 74 | 103

2. Secondary Outcome: Abstinence 3-months
Description: Report 7-day point prevalence abstinence measured at 3-months post-baseline
Time Frame: 3 months post-baseline
Population: Intention-to-treat sample
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Quitline | Specialized Quitline | Standard Quitline With Basic Needs Navigator | Specialized Quitline With Basic Needs Navigator
Number analyzed (Participants) | 485 | 485 | 484 | 490
Participants | 97 | 104 | 80 | 105

3. Secondary Outcome: 24hr Quit Attempt
Description: Report quitting smoking for at least 24 hours during intervention
Time Frame: 6 months post-baseline
Population: Intention-to-treat sample
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Quitline | Specialized Quitline | Standard Quitline With Basic Needs Navigator | Specialized Quitline With Basic Needs Navigator
Number analyzed (Participants) | 485 | 485 | 484 | 490
Participants | 241 | 219 | 248 | 235

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Standard Quitline | Specialized Quitline | Standard Quitline With Basic Needs Navigator | Specialized Quitline With Basic Needs Navigator
All-Cause Mortality (participants affected / at risk) | 0/485 | 1/485 | 1/484 | 1/490
Serious Adverse Events (participants affected / at risk) | 0/485 | 0/485 | 0/484 | 0/490
Other Adverse Events (participants affected / at risk) | 0/485 | 0/485 | 0/484 | 0/490

LIMITATIONS AND CAVEATS:
The final 9 months of the trial took place during the COVID-19 pandemic, which slowed recruitment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-03-13): https://cdn.clinicaltrials.gov/large-docs/58/NCT03194958/Prot_000.pdf
  • Statistical Analysis Plan (2017-03-08): https://cdn.clinicaltrials.gov/large-docs/58/NCT03194958/SAP_001.pdf